CLINICAL TRIAL: NCT04902716
Title: The Effectiveness of Precision Nursing Intervention Program on Cognitive Function、Sleep Quality and Emotional State of Frail Female Elderly in the Community
Brief Title: Precision Nursing Intervention Program on Cognitive Function、Sleep Quality and Emotional State of Frail Female Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Jui-Wen Yu, Master of Science, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202102EM014
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: The Effectiveness of Precision Nursing Intervention Program on Cognitive Function、Sleep Quality and Emotional State of Frail Femal Elderly in the Community
Keywords: Precision Nursing, Frail women, Cognitive function, Sleep quality, Emotional state
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Precision Nursing, Frail women, Cognitive function, Sleep quality, Emotional state, (Experimental): According to the characteristics of the elders in the community and making good use of health policies and local resources, a 12-week appropriate diversified curriculum is arranged as intervention measures.
  Interventions: Behavioral: Design course

INTERVENTIONS:
Behavioral: Design course — Precision nursing is a new trend in nursing in recent years. It is based on individual differences in disease type, gender, lifestyle, family, race, social and cultural factors, etc., to provide the most suitable empirical-based nursing treatment.Diverse courses include music, breathing exercises, cognitive training, hand-made knitting, etc.

SUMMARY:
Background: Taiwan's community population is aging rapidly, and women in the aging community account for the majority of frail elderly.In the process of aging, you must face changes in cognitive function, sleep disorders, and emotional state. Female elders have more impact on physical health than male elders. Precision nursing is a new trend in nursing in recent years. It is based on individual differences in disease type, gender, lifestyle, family, race, social and cultural factors, etc., to provide the most suitable empirical-based nursing treatment. It can also prevent and delay disability in improving the cognitive function, sleep quality and emotional state of frail female elderly in the community.

Purpose: This study explored the effectiveness of precision nursing intervention program on cognitive function,sleep quality and emotional state of frail female elderly in the community.

Methods: This study utilized a quasi-experimental research design. The subjects divided to 35 persons of experimental group and 35 people of comparison group. The experimental group implemented a weekly precision care program course for frail female elderly in the community for a total of 12 weeks; the control group maintained normal daily life. We collected cognitive function、sleep quality and emotional state from before and after intervention among frail female elderly in the community. The statistical methods uses were descriptive analysis, chi square, t test, generalized estimating equation (GEE), and difference-in-differences.

Expected benefit: The precise care plan of this study can benefit the cognitive function, sleep quality and emotional state of frail female elders in the community, and then extend it to various aging communities. According to the characteristics of the community elders and making good use of health policies and local resources, we will arrange and design appropriate courses to create a localized healthy aging life circle, and achieve the goal of preventing and delaying disability for the elderly and frail.

ELIGIBILITY:
Inclusion Criteria:

* (1) Elders over 65 years old can come and return home on their own. (2) Clear awareness and barrier-free communication. (3) Those who are frail or above detected by SOF screening, SOF ≥ 2 or above. (4) Agree to participate in this research and complete the consent form.

Exclusion Criteria:

-(1) Severe visual and hearing impairment, unable to cooperate with the researcher.

(2) Those whose limbs cannot participate in activities normally. (3) For chronic physical diseases, doctors have ordered those who are prohibited from exercising.

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Short Portable Mental State Questionnaire, SPMSQ | 1 week
  The Short Portable Mental Status Questionnaire (SPMSQ) is a widely used 10-item cognitive screening instrument,whose items test orientation to time and place, memory, current event information (date, day of the week, name of this place, telephone number, date of birth, age, name of current prime minister and previous prime minister, mother's maiden name), and calculation (subtract 3s starting with number 20). The total number of errors is computed and it ranges from 0 to 10.
Pittsburgh Sleep Quality Index, PSQI | 1 month
  The Pittsburgh Sleep Quality Index (PSQI),a self-rating questionnaire for measuring subjective sleep quality that specifically assesses the preceding I-month period . The PSQI yields a global score that is the sum of seven component scores, each of which addresses a specific aspect of subjective sleep quality.
BSRS-5 (5-item Brief Symptom Rating Scale) | 1 week
  The five items of psychological symptoms and is commonly used for screening psychological disorders and is available in Taiwan with excellent validity and reliability . For suicide prevention, the Taiwan BSRS-5 adds the sixth additional item that directly asks the subject about the urge of suicide attempts . The BSRS-5 is a 5-item, self-administered questionnaire that is derived from the 50-item brief symptom rating scale, which measures anxiety , depression , hostility , interpersonal sensitivity , and additional symptoms . The score for each item ranges from 0 to 4 (0, not at all; 1, a little bit; 2, moderately; 3, quite a bit; and 4, extremely). A total score above 14, or a score of more than 1 on the additional suicide survey item.

CONTACTS AND LOCATIONS:
Locations (1):
- Design course, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fu MR, Kurnat-Thoma E, Starkweather A, Henderson WA, Cashion AK, Williams JK, Katapodi MC, Reuter-Rice K, Hickey KT, Barcelona de Mendoza V, Calzone K, Conley YP, Anderson CM, Lyon DE, Weaver MT, Shiao PK, Constantino RE, Wung SF, Hammer MJ, Voss JG, Coleman B. Precision health: A nursing perspective. Int J Nurs Sci. 2019 Dec 24;7(1):5-12. doi: 10.1016/j.ijnss.2019.12.008. eCollection 2020 Jan 10. PMID 32099853
- [Result] Kidd T, Mold F, Jones C, Ream E, Grosvenor W, Sund-Levander M, Tingstrom P, Carey N. What are the most effective interventions to improve physical performance in pre-frail and frail adults? A systematic review of randomised control trials. BMC Geriatr. 2019 Jul 11;19(1):184. doi: 10.1186/s12877-019-1196-x. PMID 31291884
- [Result] Romera-Liebana L, Orfila F, Segura JM, Real J, Fabra ML, Moller M, Lancho S, Ramirez A, Marti N, Cullell M, Bastida N, Martinez D, Gine M, Cendros P, Bistuer A, Perez E, Fabregat MA, Foz G. Effects of a Primary Care-Based Multifactorial Intervention on Physical and Cognitive Function in Frail, Elderly Individuals: A Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2018 Nov 10;73(12):1688-1674. doi: 10.1093/gerona/glx259. PMID 29346524
- [Result] Wang WL, Chen KH, Pan YC, Yang SN, Chan YY. The effect of yoga on sleep quality and insomnia in women with sleep problems: a systematic review and meta-analysis. BMC Psychiatry. 2020 May 1;20(1):195. doi: 10.1186/s12888-020-02566-4. PMID 32357858
- [Result] Puts MTE, Toubasi S, Andrew MK, Ashe MC, Ploeg J, Atkinson E, Ayala AP, Roy A, Rodriguez Monforte M, Bergman H, McGilton K. Interventions to prevent or reduce the level of frailty in community-dwelling older adults: a scoping review of the literature and international policies. Age Ageing. 2017 May 1;46(3):383-392. doi: 10.1093/ageing/afw247. PMID 28064173